CLINICAL TRIAL: NCT02940301
Title: A Phase 2 Trial of Ibrutinib and Nivolumab in Patients With Relapsed or Refractory Classical Hodgkin's Lymphoma
Brief Title: Ibrutinib and Nivolumab in Treating Patients With Relapsed or Refractory Classical Hodgkin Lymphoma
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Responsible Party: Principal Investigator, Lapo Alinari, Principal Investigator, Ohio State University Comprehensive Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OSU-16077; NCI-2016-01473 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2016-10-18; First posted 2016-10-20 (Estimated); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Classical Hodgkin Lymphoma
MeSH Terms: interventions — ibrutinib; Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (ibrutinib, nivolumab) (Experimental): Patients receive ibrutinib PO QD on days 1-21 and nivolumab IV continuously over 60 minutes on day 1. Treatment with nivolumab repeats every 21 days for up to 16 courses and treatment with ibrutinib continues in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Ibrutinib; Other: Laboratory Biomarker Analysis; Biological: Nivolumab

INTERVENTIONS:
Drug: Ibrutinib — Given PO
  Other Names: BTK Inhibitor PCI-32765; CRA-032765; Imbruvica; PCI-32765
Other: Laboratory Biomarker Analysis — Correlative studies
Biological: Nivolumab — Given IV
  Other Names: BMS-936558; MDX-1106; NIVO; ONO-4538; Opdivo

SUMMARY:
This phase II trial studies how well ibrutinib and nivolumab work in treating patients with classical Hodgkin lymphoma that has come back or has not responded to treatment. Ibrutinib may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Monoclonal antibodies, such as nivolumab, may block cancer growth in different ways by targeting certain cells. Giving ibrutinib and nivolumab may work better in treating patients with classical Hodgkin lymphoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To estimate the complete response (CR) rate with ibrutinib at the standard dose of 560 mg daily in combination with nivolumab 3 mg/kg intravenously (IV) every 3 weeks up to 16 infusions in patients with relapsed or refractory classical Hodgkin lymphoma (cHL).

SECONDARY OBJECTIVES:

I. To determine the overall response rate (ORR) with ibrutinib and nivolumab in combination in patients with relapsed or refractory classical HL.

II. To determine safety and toxicity of ibrutinib in combination with nivolumab in patients with relapsed or refractory cHL.

III. To determine the progression free survival (PFS) in patients with relapsed or refractory cHL treated with combined ibrutinib and nivolumab.

IV. To determine the duration of response in patients with relapsed or refractory cHL treated with ibrutinib in combination with nivolumab.

TERTIARY OBJECTIVES:

I. To determine the effects of ibrutinib and nivolumab on the distribution of T-, B-, and NK cells in the peripheral blood.

II. To determine the effects of ibrutinib and nivolumab on Th1/Th2 cytokines profile and correlate this with treatment response.

III. To determine the effects of ibrutinib and nivolumab on Th1/Th2 ration and specific IgG sub-isotypes.

OUTLINE:

Patients receive ibrutinib orally (PO) once daily (QD) on days 1-21 and nivolumab IV continuously over 60 minutes on day 1.Treatment with nivolumab repeats every 21 days for up to 16 courses and treatment with ibrutinib continues in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up periodically.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically confirmed classical HL that is relapsed or refractory after at least one prior therapy are eligible

  * Patients with lymphocyte predominant Hodgkin's are eligible
* Prior treatments: patients must have had at least one prior therapy

  * Patients with previous autologous transplant are permitted
  * Patients who are eligible and willing to undergo autologous transplant should not be enrolled on this trial
  * Prior allogeneic transplant is NOT permitted
  * Prior treatment with Bruton's tyrosine kinase (BTK) inhibitors is NOT permitted
  * Prior treatment with nivolumab is permitted
* Presence of radiographically measurable disease (defined as the presence of a >= 1.0 cm lesion, as measured in the longest dimension by computed tomography [CT] scan or positron emission tomography [PET]/CT scan or magnetic resonance imaging [MRI] scan)
* Absolute neutrophil count (ANC) > 1000/uL
* Platelets > 75,000/uL
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) =< 2 x upper limit of normal (ULN)
* Total bilirubin =< 1.5 x ULN
* Creatinine =< 2.0 mg/dl
* Eastern Cooperative Oncology Group (ECOG) performance status of =< 2
* Patients with human immunodeficiency virus (HIV) are not permitted to enroll
* Patients with history of hepatitis B or C infection are not permitted to enroll; to enroll patients must have no evidence of hepatitis B or C surface antigen (Ag) and negative hepatitis B core antibody (Ab); patients previously immunized for hepatitis B who are hepatitis B surface Ab positive, but surface Ag and core Ab negative are eligible
* Non-pregnant and non-nursing; pregnant and nursing patients may not be enrolled; women and men of reproductive potential must agree to use acceptable forms of contraception during the study
* Willing and able to participate in all required evaluations and procedures in this study protocol including swallowing capsules without difficulty
* Ability to understand the purpose and risks of the study and provide signed and dated informed consent and authorization to use protected health information (in accordance with national and local subject privacy regulations)

Exclusion Criteria:

* Prior malignancy, except for adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, or other cancer from which the subject has been disease free for >= 2 years or which will not limit survival to < 2 years
* A life-threatening illness, medical condition or organ system dysfunction which, in the investigator's opinion, could compromise the subject's safety, interfere with the absorption or metabolism of ibrutinib, or put the study outcomes at undue risk
* Significant cardiovascular disease such as uncontrolled or symptomatic arrhythmias, congestive heart failure, or myocardial infarction within 6 months of screening, or any class 3 or 4 cardiac disease as defined by the New York Heart Association Functional Classification
* Malabsorption syndrome, disease significantly affecting gastrointestinal function, or resection of the stomach or small bowel, symptomatic inflammatory bowel disease, partial or complete bowel obstruction, or gastric restrictions and bariatric surgery, such as gastric bypass
* Central nervous system (CNS) involvement by lymphoma
* Has a diagnosis of immunosuppression or is receiving ongoing immunosuppressive therapy, including systemic or enteric corticosteroids for treatment of lymphoid cancer or other conditions

  * Note: subjects may use topical or inhaled corticosteroids or low-dose steroids (=< 20 mg of prednisone or equivalent per day) as therapy for comorbid conditions; during study participation, subjects may also receive systemic or enteric corticosteroids as needed for treatment-related toxicities
* Has an active autoimmune disease or history of autoimmune disease such as hepatitis, hypophysitis, nephritis, hyperthyroidism or hypothyroidism, interstitial lung disease, colitis
* Requires or is currently receiving anticoagulation with warfarin or equivalent vitamin K antagonists (eg, phenprocoumon) within 28 days of first dose of study drug
* Requires treatment with a strong cytochrome P450 (CYP) 3A inhibitor
* Currently active, clinically significant hepatic impairment Child-Pugh class B or C according to the Child Pugh classification
* Major surgery within 4 weeks before first dose of study drug
* History of stroke or intracranial hemorrhage within 6 months before the first dose of study drug

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2016-12-20 (Actual); Primary Completion 2026-01-15 (Estimated); Study Completion 2026-02-15 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients in CR | Up to course 7 (147 days)
  Simon's two-stage design will be used to test the null hypothesis that the true CR rate is =< 20% versus the alternative hypothesis that the true CR rate is >= 50%.

SECONDARY OUTCOMES:
Duration of response | From the first documentation of response (CR, partial response) to the first documentation of definitive disease progression or death from any cause, whichever occurs first, assessed up to 3 years
  Kaplan-Meier methods will be used to estimate duration of response curves and corresponding quantiles (including the median).
Incidence of adverse events measured by Common Terminology Criteria for Adverse Events version 4.03 | Up to 3 years
  Will be summarized by type and grade, including incidence of grade 3+ adverse events. Initially, adverse event data will be summarized regardless of attribution, but may also be summarized for treatment-related adverse events. Number of cycles administered and reasons for treatment discontinuation will also be summarized to assess tolerability.
ORR | Up to 3 years
  Defined as the number of patients who achieve a complete or partial remission divided by the number of evaluable patients, will be calculated with an exact 90% confidence interval.
PFS | From the date of enrollment until the first documentation of objective disease progression or death from any cause, whichever occurs first, assessed up to 3 years
  Kaplan-Meier methods will be used to estimate the PFS curves and corresponding quantiles (including the median).

CONTACTS AND LOCATIONS:
Overall Officials: Lapo Alinari, MD, PhD, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (2):
- United States (2):
  - Winship Cancer Center of Emory University, Atlanta, Georgia
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Jamesline — http://cancer.osu.edu